Project Title: Effects of transcranial direct current stimulation (tDCS) on cognition in older adults with mild cognitive impairment: A randomized controlled trial

Date of document: June 6, 2022



Project Title: Effects of transcranial direct current stimulation (tDCS) on cognition in older adults with mild cognitive impairment: A randomized controlled trial

Principle Investigator: Dr. Michael KUO Associate Professor of Tung Wah College

Participant:

The study was initiated by the School of Medical and Health Sciences of Tung Wah College. We sincerely invite you to participate in a research activity on transcranial direct current stimulation (tDCS). If you agree, we will conduct one interview session, three 90-minute cognitive assessment sessions, and 8 20-minute tDCS sessions. Before each assessment session, we will put a cap on for you. After that, you need to complete computerized memory tasks. Your EEG will be collected by the cap while you do the memory tasks.tDCS may cause a slight tingling and itching sensation. However, this study will not pose any danger to the participants. The entire training aims to study the effects of tDCS on memory in older adults with memory impairment potentially. It will help rehabilitation professionals to understand whether tDCS can help to improve their memory.

I guarantee that all your personal data will be kept strictly confidential. Records are kept with passwords to ensure the security of the data. The results of the research will be published in appropriate academic conferences and journals, and your personal identity will not be disclosed or identified in the relevant reports. The research data will be retained after the deletion of personal data for future comparative analysis of other research data. If you have any comments, please contact Dr. Michael KUO (office number 3468 6656 or email michaelkuo@twc.edu.hk). If you have any complaints about the researchers, you can contact the Research Office of Tung Wah College (Office Tel: 3190 6686). Thank you for your support.